CLINICAL TRIAL: NCT00989027
Title: Impact of Uterotonic Agents on Isolated Human Myometrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-08
Record Dates: First submitted 2009-07-29; First posted 2009-10-02 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Dose-response; Oxytocin pre-treatment
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Ergonovine; Carboprost; carboprost tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No treatment (No Intervention): A control sample from each patient (no uterotonic drug applied) will be measured concurrently with samples treated with various drugs.
- Treatment (Active Comparator): Samples from each patient will be bathed in solutions containing varying concentrations of either oxytocin, carboprost and ergonovine, and contractility will be measured.
  Interventions: Drug: Oxytocin; Drug: Ergonovine; Drug: Carboprost; Drug: Oxytocin and Ergonovine; Drug: Oxytocin and Carboprost

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 10-9mol/L to 10-3mol/L, in Krebs-Henseleit solution.
  Arms: Treatment
Drug: Ergonovine — Ergonovine, 10-9mol/L to 10-3mol/L, in Krebs-Henseleit solution.
  Other Names: Ergonovine Maleate
  Arms: Treatment
Drug: Carboprost — Carboprost, 10-9mol/L to 10-3mol/L, in Krebs-Henseleit solution.
  Other Names: Hemabate
  Arms: Treatment
Drug: Oxytocin and Ergonovine — Oxytocin and Ergonovine, 10-9mol/L to 10-3mol/L, in Krebs-Henseleit solution.
  Other Names: Oxytocin; Ergonovine
  Arms: Treatment
Drug: Oxytocin and Carboprost — Oxytocin and Carboprost, 10-9mol/L to 10-3mol/L, in Krebs-Henseleit solution.
  Other Names: Oxytocin; Hemabate
  Arms: Treatment

SUMMARY:
The purpose of this study is to compare the ability of a sample of uterine muscle tissue to contract in the presence of various drugs. The drugs studied are typically used to contract the uterus when a pregnant patient continues to bleed after delivery. Amongst the uterotonic drugs (used to contract the uterus), namely oxytocin, ergonovine and carboprost, the most effective one to use is not known.

The investigators will be testing uterine muscle samples in the presence of these drugs at various concentrations, to see what their contractility measures over time, as compared with a control sample, in which no drugs will be applied.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a major cause of maternal mortality and morbidity. In 80% cases of PPH, the primary cause is failure of the uterus to contract after delivery of the baby, which then requires further treatment of the mother with uterotonic drugs (drugs used to contract uterus and thus prevent bleeding).

Patients participating in this study will be asked to donate a very small sample of uterine tissue during Cesarean section, which will be tested for the ability to contract after treatment with various uterotonic drugs (oxytocin, ergonovine and carboprost) in the laboratory. This information will help us know the effect of these drugs by comparing the contractile capability of the uterine tissue.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary Cesarean section
* Cesarean section under spinal anesthesia

Exclusion Criteria:

* Patients who require general anesthesia
* Patient who had previous uterine surgery or Cesarean section
* Patients with placental anomalies
* Emergency Cesarean section in labor
* Patients with bleeding disorders

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Amplitude of contraction | 6-8 hours

SECONDARY OUTCOMES:
Integrated area under response curve (AUC) | 6-8 hours
Basal tone | 6-8 hours
Frequency of contraction | 6-8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada